CLINICAL TRIAL: NCT01347762
Title: Nabilone for Cannabis Dependence: A Pilot Study
Acronym: NAB CAN
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kevin P. Hill, MD, MHS, Psychiatrist-In-Charge, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010-P-000096; 1K99DA029115-01 (NIH)
Record Dates: First submitted 2011-04-26; First posted 2011-05-04 (Estimated); Results first posted 2018-06-01 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Cannabis Dependence; Marijuana Dependence
Keywords: cannabis dependence; marijuana dependence; cannabis use disorders; cannabis withdrawal; nabilone
MeSH Terms: conditions — Marijuana Abuse | interventions — nabilone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nabilone (Experimental): nabilone titrated to 2 mg daily
  Interventions: Drug: Nabilone
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nabilone — nabilone titrated to 1 mg by mouth twice daily
  Other Names: Nabilone (Cesamet), CSA Drug Code 7379, Schedule II, NDC 0037-1221-50
  Arms: Nabilone
Drug: Placebo — one placebo capsule by mouth twice daily
  Arms: Placebo

SUMMARY:
Cannabis use disorders are an important public health problem in the United States, but there are no effective medications available to treat these disorders. The investigators intend to test a medication with interesting properties, nabilone, as a treatment for cannabis dependence and to study the relationship of this treatment with the brain using functional MRI brain scans. Nabilone and marijuana have similar effects upon behaviors and the human body, suggesting that nabilone may decrease cannabis withdrawal symptoms while allowing treatment-seeking patients to benefit from behavioral treatments when they are trying to stop using cannabis. The investigators propose to assess the relationship of nabilone, when added to behavioral treatment, on cannabis use patterns in cannabis-dependent patients. The investigators also aim to determine the effects of nabilone on performance on neuropsychological tests and to assess the correlation of neuropsychological performance to brain changes using functional MRI brain scans. The investigators hypothesize that patients receiving nabilone will reduce their use of cannabis more than patients receiving placebo during this 10-week treatment trial.

DETAILED DESCRIPTION:
Cannabis use disorders are an important public health problem in the United States, but no effective pharmacotherapies are available to treat these disorders. The investigators intend to test a novel agonist pharmacotherapy, nabilone, for cannabis dependence and to study the relationship of this treatment with the brain using BOLD fMRI measures. The behavioral and physiological effects of nabilone and Δ9-THC overlap, suggesting that nabilone may ameliorate cannabis withdrawal symptoms while allowing treatment-seeking outpatients to benefit from medical management (MM) sessions when they are trying to stop using cannabis. The investigators propose to assess the relationship of nabilone, when added to MM, on cannabis use patterns in cannabis-dependent patients. The investigators also aim to determine the effects of nabilone on performance on neuropsychological tests and to assess the correlation of neuropsychological performance to brain changes using BOLD fMRI measures.

In this pilot study, subjects will receive either nabilone or placebo in addition to medical management (MM) over a 10-week treatment period. Subjects' responses to neuropsychological testing carried out while the subject is receiving fMRI scans at 3 time points: at baseline, 4 weeks, and 10 weeks. Following treatment completion, subjects will have a follow-up visit at 14 weeks. This pilot study will evaluate the feasibility of nabilone treatment for cannabis dependence and will establish effect sizes for a larger trial in which subjects will receive high-dose nabilone, low-dose nabilone, or placebo in addition to MM.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-45 years
* DSM-IV diagnosis of cannabis dependence, based on the Structured Clinical Interview for DSM-IV (SCID)
* express a desire to quit cannabis use within the next 30 days
* have used cannabis on more than4 days within the past 30 days
* for women of childbearing age, a negative pregnancy test at screening with agreement to use adequate contraception to prevent pregnancy and monthly pregnancy tests
* consent for us to communicate with their prescribing clinician
* furnish the names of 2 locators, who would assist study staff in locating them during the study period
* live close enough to McLean Hospital to attend study visits
* plan to stay in the Boston area for the next 3 months
* are willing and able to sign informed consent.

Exclusion Criteria:

* current diagnosis of other drug or alcohol dependence (excluding nicotine)
* recent (within 3 months) significant cardiac disease
* current serious psychiatric illness or history of psychosis, schizophrenia, bipolar type I disorder
* current medical condition (including significant laboratory abnormalities, such as liver function tests >5 times the upper limit of normal range) that could prevent regular study attendance
* mental retardation or organic mental disorder
* acutely dangerous or suicidal behavior
* currently in a residential treatment setting in which substance use is monitored and restricted, since the restricted access to drugs could represent an important confounding variable
* pregnant, nursing, or, if a woman of childbearing potential, not using a form of birth control judged by the investigator to be effective
* concomitant daily treatment with opioid analgesics, sedative hypnotics, or other known CNS depressants
* known hypersensitivity to cannabinoids or sesame oil
* disease of the gastrointestinal system, liver, or kidneys that may impede metabolism or excretion of nabilone
* inability to read or write in English. The potential hazards of a Schedule II medication like nabilone underscore the importance of English proficiency in this medication trial.
* unwilling or unable to participate in MRI scanning (e.g., those having pacemakers, bone plates, screws, etc.; claustrophobia)
* a history of seizures, head trauma or other history of CNS insult that could predispose the subject to seizures .

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2010-06; Primary Completion 2017-06-09 (Actual); Study Completion 2017-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin P Hill, MD, MHS, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 14 potential subjects were screened but did not qualify for Phase 1 and 18 for Phase 2. Reasons included: positive urine screen for opiates or cocaine, lost to follow up after screening visit, withdrew from the study due to time constraints before randomization, met criteria for alcohol dependence or did not test positive for THC urine screen
Groups:
- Nabilone Titrated 2 mg Daily (Phase 1): nabilone titrated to 2 mg daily
  Nabilone: nabilone titrated to 1 mg by mouth twice daily
- Placebo (Phase 1); Placebo (Phase 2): Placebo
  Placebo: one placebo capsule by mouth twice daily
- Nabilone Titrated to 4 mg Daily (Phase 2): nabilone titrated to 4 mg daily
  Nabilone: nabilone titrated to 2 mg by mouth twice daily
Period: Overall Study
Arm/Group | Nabilone Titrated 2 mg Daily (Phase 1) | Placebo (Phase 1) | Nabilone Titrated to 4 mg Daily (Phase 2) | Placebo (Phase 2)
Started | 10 | 8 | 16 | 18
Completed | 6 | 6 | 7 | 10
Not Completed | 4 | 2 | 9 | 8
Not completed — Lost to Follow-up | 0 | 1 | 6 | 5
Not completed — Withdrawal by Subject | 4 | 1 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nabilone Titrated 2 mg Daily (Phase 1) | Placebo (Phase 1) | Nabilone Titrated to 4 mg Daily (Phase 2) | Placebo (Phase 2) | Total
Number analyzed (Participants) | 10 | 8 | 16 | 18 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.40 (5.17) | 28.88 (7.53) | 27.81 (6.81) | 28.11 (7.26) | 27.42 (6.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 11 | 11 | 28
  Male | 7 | 5 | 5 | 7 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 6 | 2 | 13
  White | 6 | 6 | 9 | 15 | 36
  More than one race | 1 | 0 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Baseline Urine THC/Creatinine Ratio [Mean (Standard Deviation); unit: Ratio] | 491.6 (283.0) | 458.7 (568.9) | 633.2 (728.5) | 371.0 (265.4) | 489.8 (496.1)
Average Number of Inhales of Marijuana Per Day [Mean (Standard Deviation); unit: Inhales per day] | 50.1 (43.8) | 27.1 (13.2) | 28.9 (31.8) | 16.53 (29.13) | 30.52 (33.65)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Cannabis Use at 10 Weeks
Description: Quantitative cannabis urine screens (THC-COOH:Creatinine ratio)
Time Frame: baseline and 10 weeks
Population: Fewer participants had their THC:creatinine ratios analyzed than were randomized due to a high number of subject drop-out. Any subject who dropped out before completing the 10 weeks of treatment were not analyzed using this measure.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Nabilone Titrated 2 mg Daily (Phase 1) | Placebo (Phase 1) | Nabilone Titrated to 4 mg Daily (Phase 2) | Placebo (Phase 2)
Number analyzed (Participants) | 6 | 6 | 8 | 10
Ratio | 268.8 (183.0) | 286.7 (349.7) | 490.3 (615.0) | 216.9 (188.5)

2. Primary Outcome: Number of Marijuana Inhales Per Day
Description: Average # of marijuana inhales per day during baseline compared to after 10 weeks of treatment.
Time Frame: Week 10
Population: Fewer participants had their "average number of inhales per day" analyzed than were randomized due to a high number of subject drop-out. Any subject who dropped out before completing the 10 weeks of treatment were not analyzed using this measure.
Measure: Mean (Standard Deviation); unit: Inhales per day
Arm/Group | Nabilone Titrated 2 mg Daily (Phase 1) | Placebo (Phase 1) | Nabilone Titrated to 4 mg Daily (Phase 2) | Placebo (Phase 2)
Number analyzed (Participants) | 6 | 6 | 8 | 10
Inhales per day | 33.8 (31.0) | 22.6 (30.6) | 15.8 (35.6) | 10.6 (14.6)

3. Secondary Outcome: Change From Baseline Neuropsychological Performance at 4 Weeks
Description: performance on neuropsychological tests administered inside of the fMRI scanner and outside of the fMRI scanner
Time Frame: baseline and 4 weeks
Population: Due to funding and the principal investigator's change in institutions, this data was not analyzed and is no longer available to the investigator.
Arm/Group | Nabilone Titrated 2 mg Daily (Phase 1) | Placebo (Phase 1) | Nabilone Titrated to 4 mg Daily (Phase 2) | Placebo (Phase 2)
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline Cannabis Use at 14 Weeks
Description: quantitative urine screens - Comparing the THC-COOH to creatinine ratio at baseline and at the end of the study (Week 14)
Time Frame: baseline and 14 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Nabilone Titrated 2 mg Daily (Phase 1) | Placebo (Phase 1) | Nabilone Titrated to 4 mg Daily (Phase 2) | Placebo (Phase 2)
Number analyzed (Participants) | 6 | 6 | 8 | 10
Ratio | 524.2 (466.2) | 326.7 (403.7) | 297.7 (291.8) | 222 (186.53)

5. Secondary Outcome: Change From Baseline in Neuropsychological Performance at 10 Weeks
Description: performance on neuropsychological tests administered inside of the fMRI scanner and outside of the fMRI scanner
Time Frame: baseline and 10 weeks
Population: as for outcome 3
Arm/Group | Nabilone Titrated 2 mg Daily (Phase 1) | Placebo (Phase 1) | Nabilone Titrated to 4 mg Daily (Phase 2) | Placebo (Phase 2)
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time the subject was randomized up until the subject's last visit, this encompasses a total of 14 weeks per subject.
Description: During every visit (twice a week) a study staff member would ask the subject if they were experiencing any adverse events from the medication or participation in the study. Furthermore, during the weekly medication management session with the study physician, the physician asked and checked for adverse events as well
Arm/Group | Nabilone Titrated 2 mg Daily (Phase 1) | Placebo (Phase 1) | Nabilone Titrated to 4 mg Daily (Phase 2) | Placebo (Phase 2)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8 | 0/16 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8 | 0/16 | 0/18
Other Adverse Events (participants affected / at risk) | 0/10 | 0/8 | 0/16 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-14): https://cdn.clinicaltrials.gov/large-docs/62/NCT01347762/Prot_SAP_000.pdf